CLINICAL TRIAL: NCT05722899
Title: Ten Weeks of Recreational Football Training in 55- to 70-year-old Adults: Effects on Muscle Power, Functional Capacity, Body Composition and Endurance Exercise Capacity
Brief Title: Football 4 Health in Middle-aged to Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Evelien Van Roie, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S64926
Record Dates: First submitted 2023-01-20; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Exercise Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Football training (Experimental): 10-week football training program with small-sided games, 2x/week, 45min-1h
  Interventions: Other: Football training
- Control (No Intervention): No intervention, no changes in lifestyle and diet

INTERVENTIONS:
Other: Football training — 10-week progressive football training with small-sided games, 2x/week, 45min-1h sessions
  Arms: Football training

SUMMARY:
Ageing in humans is accompanied by a progressive decline in lower-limb muscle power production. In addition to a decline in musculoskeletal fitness, ageing is associated with a reduction in cardiovascular and metabolic fitness. Therefore, if exercise interventions aim for a high impact on the overall health status of middle-aged and older adults, they should combine endurance, high-intensity interval training and muscular strengthening activities. Recreational football training combines all these training components, which implies that it could constitute an adequate training modality for participants of all ages. What remains to be investigated in more detail, is whether recreational football training can improve muscle power production in middle-aged to older adults and whether this potential improvement is present across the full force-velocity (F-V) profile. Next to a detailed analysis of the leg-extensor F-V profile as primary outcome, simultaneous effects on functional capacity, body composition and endurance exercise capacity were investigated. In addition, feasibility and the physical demands (internal and external load indicators) of the training program were tracked throughout the intervention period.

ELIGIBILITY:
Exclusion Criteria:

* Unstable cardiovascular disease
* Neurological disorders
* Cognitive malfunctioning
* Acute infections or fever
* Severe musculoskeletal problems
* Systematic engagement in (resistance) exercise in the 12 months prior to participation

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Maximal power | Time Frame: Change from baseline in maximal power (watt) at 12 weeks
  Force-velocity profiling is carried out unilaterally (dominant leg) on the pneumatic leg press device (Leg Press CC, HUR, Kokkola, Finland). The test protocol consists of a maximal isometric test (knee joint angle = 85°, hip angle = 55°; 3 attempts of 3s), followed by explosive concentric leg extensions at gradually increasing loads (unloaded, 15%, 30%, 45%, 60%, 75% of the maximal isometric force, 2-3 attempts per load, and additional single repetitions until one-repetition maximum is reached). Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced adaptations. Maximal power is used for the analyses.
Maximal force | Time Frame: Change from baseline in maximal force (N) at 12 weeks
  Force-velocity profiling is carried out unilaterally (dominant leg) on the pneumatic leg press device (Leg Press CC, HUR, Kokkola, Finland). The test protocol consists of a maximal isometric test (knee joint angle = 85°, hip angle = 55°; 3 attempts of 3s), followed by explosive concentric leg extensions at gradually increasing loads (unloaded, 15%, 30%, 45%, 60%, 75% of the maximal isometric force, 2-3 attempts per load, and additional single repetitions until one-repetition maximum is reached). Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced adaptations. Maximal force is used for the analyses.
Maximal velocity | Time Frame: Change from baseline in maximal velocity (m/s) at 12 weeks
  Force-velocity profiling is carried out unilaterally (dominant leg) on the pneumatic leg press device (Leg Press CC, HUR, Kokkola, Finland). The test protocol consists of a maximal isometric test (knee joint angle = 85°, hip angle = 55°; 3 attempts of 3s), followed by explosive concentric leg extensions at gradually increasing loads (unloaded, 15%, 30%, 45%, 60%, 75% of the maximal isometric force, 2-3 attempts per load, and additional single repetitions until one-repetition maximum is reached). Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced adaptations. Maximal velocity is used for the analyses.
Slope of F-V profile | Time Frame: Change from baseline in the slope of F-V profile at 12 weeks
  Force-velocity profiling is carried out unilaterally (dominant leg) on the pneumatic leg press device (Leg Press CC, HUR, Kokkola, Finland). The test protocol consists of a maximal isometric test (knee joint angle = 85°, hip angle = 55°; 3 attempts of 3s), followed by explosive concentric leg extensions at gradually increasing loads (unloaded, 15%, 30%, 45%, 60%, 75% of the maximal isometric force, 2-3 attempts per load, and additional single repetitions until one-repetition maximum is reached). Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced adaptations. The equation's slope is used for the analyses.

SECONDARY OUTCOMES:
Exercise adherence | Total adherence over 10-week period
  Number of sessions attended as a percentage of total sessions planned
Enjoyment | within 1 week post-intervention
  Question: 'How much did you enjoy the training program?' Answer: 11-point Likert scale (0 = 'not at all...' to 10 = 'very...'
Score on feasibility questionnaire | within 1 week post-intervention
  Question: 'How feasible was the training program for you?' Answer: 11-point Likert scale (0 = 'not at all...' to 10 = 'very...'
Future intention to participate | within 1 week post-intervention
  Question: 'How high is the chance that you subscribe for a new sequence of training sessions?' Answer: 11-point Likert scale (0 = 'not at all...' to 10 = 'very...'
External load: total distance | Average calculated over 10-week period
  Total distance covered per training session, measured by means of GPS metrics
External load: meters in speed zones | Average calculated over 10-week period
  Total meters in different speed zones per training session, measured by means of GPS metrics
Internal load: time in speed zones | Average calculated over 10-week period
  Total time in different speed zones per training session, measured by means of GPS metrics
External load: number of accelerations | Average calculated over 10-week period
  Number of accelerations (> 2m/s²), measured by means of GPS metrics
External load: number of decelerations | Average calculated over 10-week period
  Number of decelerations (< -2m/s²), measured by means of GPS metrics
Internal load: average heart rate | Average calculated over 10-week period
  Average heart rate (percent of heart rate max) during training session, measured by means of heart rate sensor
Internal load: time in heart rate zone | Average calculated over 10-week period
  Total time in different heart rate zones per training session, measured by means of heart rate sensor
Gait speed | Change from baseline in gait speed at 10 weeks
  The average speed to walk 10m as fast as possible (in m/s)
Countermovement jump height | Change from baseline in countermovement jump height at 10 weeks
  Jump height (cm) in a countermovement jump
Timed up and go | Change from baseline in timed up and go time at 10 weeks
  Time (in s) needed to stand up from a chair, walk 3 m, turn, walk back and sit down again (as fast as possible)
5-repetition sit-to-stand time | Change from baseline in sit-to-stand performance at 10 weeks
  The time (s) needed to perform 5 sit-to-stand transitions.
5-repetition sit-to-stand power | Change from baseline in sit-to-stand performance at 10 weeks
  The power (watt) needed to perform 5 sit-to-stand transitions.
Stair ascent time | Change from baseline in stair climbing performance at 10 weeks
  The time (s) needed to ascend a flight of stairs.
Stair ascent power | Change from baseline in stair climbing performance at 10 weeks
  The power (watt) needed to ascend a flight of stairs.
Body fat percentage | Change from baseline in body fat percentage at 10 weeks
  Percentage of body fat, measured with bio-electrical impedance analysis
Skeletal muscle mass | Change from baseline in skeletal muscle mass at 10 weeks
  Skeletal muscle mass, estimated with bio-electrical impedance analysis
Running speed at 2mM lactate | Change from baseline in running speed at 10 weeks
  Endurance exercise capacity test on treadmill: running speed at 2mM lactate value
Running speed at 4mM lactate | Change from baseline in running speed at 10 weeks
  Endurance exercise capacity test on treadmill: running speed at 4mM lactate value
Rate of perceived exertion (RPE) | Change from baseline in RPE at 10 weeks
  RPE of the common highest intensity block, completed in the pre- as well as post-intervention test (i.e., values at the same speed level in both tests)
Lactate value | Change from baseline in lactate at 10 weeks
  Lactate value of the common highest intensity block, completed in the pre- as well as post-intervention test (i.e., values at the same speed level in both tests)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Movement Sciences, Leuven, Belgium